CLINICAL TRIAL: NCT05411146
Title: A Phase 1, Open-label Study to Assess the Absorption, Metabolism, and Excretion, Including the Mass Balance, of a Single Oral Dose of [14C]-Etrumadenant in Healthy Male Subjects
Brief Title: A Study Investigating the Safety, Absorption, and Elimination of Radioactively Labeled Etrumadenant, a New Compound in the Treatment of Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ARC-19; 2022-000822-50 (EudraCT Number)
Record Dates: First submitted 2022-05-10; First posted 2022-06-09 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Healthy Participants
Keywords: Etrumadenant; Pharmacokinetics; AB928; Healthy participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-etrumadenant (Experimental): Participants will receive a single dose of [14C]-etrumadenant.
  Interventions: Drug: [14C]-etrumadenant

INTERVENTIONS:
Drug: [14C]-etrumadenant — Administered as specified in the treatment arm.
  Other Names: [14C]-AB928

SUMMARY:
This study will assess absorption, metabolism, and excretion of Radioactively Labeled Etrumadenant in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.0 to 32.0 kg/m2
* Body weight ≥50 kg
* Good physical and mental health on the basis of medical history, physical examination, clinical laboratory, ECG, and vital signs, as judged by the Investigator.
* All clinical laboratory test results within the normal range or showing no clinically relevant deviations as judged by the Investigator.
* Male subjects, if not surgically sterilized, must agree to use adequate contraception and not donate sperm from (first) admission to the clinical research center until 90 days after the study drug administration. Adequate contraception for the male subject (and his female partner, if she is of childbearing potential) is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm, a cervical cap, or a condom. Total abstinence from heterosexual intercourse, in accordance with the lifestyle of the subject, is also acceptable.

Exclusion Criteria:

* Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol) at screening or admission to the clinical research center.
* Significant and/or acute illness within 5 days prior to drug administration that may impact safety assessments, in the opinion of the Investigator.
* Irregular defecation pattern (less than once per 2 days).
* For a study with a radiation burden of superior to 0.1 mSv, the subject will be excluded if he participated in another study with a radiation burden of superior to 0.1 mSv and inferior or equal to 1 mSv in the period of 1 year prior to screening; a radiation burden of superior to 1.1 mSv and inferior or equal 2 mSv in the period of 2 years prior to screening; a radiation burden of superior to 2.1 mSv and inferior or equal 3 mSv in the period of 3 years prior to screening.
* Exposure to radiation for diagnostic reasons (except dental X rays and plain X rays of thorax and bony skeleton [excluding spinal column]), during work, or during participation in a clinical study in the period of 1 year prior to screening.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Excretion of total radioactivity in urine | Up to 25 days
Excretion of total radioactivity in feces | Up to 25 days
Percentage of total radioactivity in urine at selected time points | Up to 25 days
Percentage of total radioactivity in feces at selected time points | Up to 25 days
Mass balance recovery of total radioactivity in urine | Up to 25 days
Mass balance recovery of total radioactivy in feces | Up to 25 days
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to 38 days
Number of participants with abnormal electrocardiogram (ECG) readings, abnormal vital signs, abnormal physical examinations and abnormal clinical laboratory tests results | Up to 38 days

SECONDARY OUTCOMES:
Percentage of total radioactivity in blood | Up to 24 days
Percentage of total radioactivity in plasma | Up to 24 days
Maximum Observed Plasma Concentration (Cmax) | Up to 25 days
Time to Cmax (Tmax) | Up to 25 days
Area Under the Curve From 0 to Last Observed Non-zero Concentration (AUC [0-Last]) | Up to 25 days
Area Under the Curve From Time '0' Extrapolated to Infinity (AUC[0-inf]) | Up to 25 days
Elimination Half-life (t1/2) | Up to 25 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (1):
- PRA Health Sciences (PRA) - Early Development Services (EDS), Groningen, NZ, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-19 - Lay Summary (English Version) — https://trials.arcusbio.com/study/?id=ARC-19